CLINICAL TRIAL: NCT01116687
Title: A Phase 2 Open-Label Study of RO4929097 in Metastatic Colorectal Cancer
Brief Title: RO4929097 in Treating Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02845; NCI-2012-02845 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MCC 16221 (Other: H. Lee Moffitt Cancer Center and Research Institute); 8537 (Other: CTEP); N01CM62208 (NIH); P30CA076292 (NIH)
Record Dates: First submitted 2010-04-28; First posted 2010-05-05 (Estimated); Results first posted 2012-06-11 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2012-12

CONDITIONS: Recurrent Colon Cancer; Recurrent Rectal Cancer; Stage IV Colon Cancer; Stage IV Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — 2,2-dimethyl-N-(6-oxo-6,7-dihydro-5H-dibenzo(b,d)azepin-7-yl)-N'-(2,2,3,3,3-pentafluoropropyl)malonamide

ARMS (1):
- Treatment (RO4929097) (Experimental): See detailed description.
  Interventions: Drug: gamma-secretase/Notch signalling pathway inhibitor RO4929097; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: gamma-secretase/Notch signalling pathway inhibitor RO4929097 — Given orally
  Other Names: R4733; RO4929097
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial studies how well RO4929097 works in treating patients with metastatic colorectal cancer. RO4929097 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the objective radiographic response rate associated with RO4929097 in patients with metastatic colorectal cancer who have progressed following at least two prior treatments in the metastatic setting.

SECONDARY OBJECTIVES:

I. To determine the progression-free survival (PFS) and overall survival (OS) associated with this agent.

II. To determine the safety and tolerability of RO4929097 in this patient population.

III. To assess whether response correlates with up regulation of the Notch pathway, to be determined through immunohistochemical analysis of Notch1, ICN and HES1 on available paraffin-embedded tissue samples (exploratory aim).

OUTLINE:

Participants will take 20 mg of RO4929097 by mouth at home in the morning for 3 days and then not take it for 4 days, continuously. The tablet is to be taken at approximately the same time the days they take it on an empty stomach, 1 hour before a meal or 2 hours after a meal. Participants will be asked to keep a "pill diary" recording each dose of study drug (including missed, skipped, or vomited doses) and return the diary to the study staff each visit. Participants will be informed that tablets should not be broken or opened; that they should avoid eating grapefruits or drinking grapefruit juice while on the study; that if they miss a dose of study drug, they should not try to make up that dose; that instead, they should wait until their next scheduled dose. Participants will see their study doctor and undergo standard blood work (approximately 12 mL) every 4 weeks. During these visits, participants will be asked about side effects of the RO4929097 and undergo a physical examination. Participants will continue taking the RO4929097 as long as they are tolerating it and as long as the cancer is shrinking or remains stable.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed colorectal cancer (NOS 10010029) with evidence of stage 4 disease (distant metastases)
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm with conventional techniques or as >= 10 mm with spiral CT scan
* Patients must have received at least two prior lines of treatment in the metastatic setting; patients must have received 5-Fluorouracil (5-FU) or capecitabine, oxaliplatin and irinotecan, either in the adjuvant or metastatic setting; at least 4 weeks must have elapsed since prior chemotherapy or radiation therapy (6 weeks if the last regimen included mitomycin C)
* Life expectancy of greater than 3 months
* ECOG performance status =<2 (Karnofsky >= 60%)
* Absolute neutrophil count >= 1,000/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 9 g/dL
* Total bilirubin =< 1.5 x institutional upper limit of normal
* AST(SGOT)/ALT(SGPT) =< 2.5 x institutional upper limit of normal (or =< 5 x institutional upper limit of normal in patients with liver metastases)
* Creatinine =< 1.5 x institutional upper limit of normal
* The effects of RO4929097 on the developing human fetus at the recommended therapeutic dose are unknown; Notch signal pathway inhibitors are known to cause interruption of the embryonic signaling pathway and may lead to serious or life-threatening birth defects, including brain deformities, facial malformation, heart problems, or abnormal organs; therefore, women of childbearing potential and men must use two forms of contraception (i.e., barrier contraception and one other method of contraception) at least 4 weeks prior to study entry, for the duration of study participation, and for at least 3 months post-treatment; should a woman become pregnant or suspect she is pregnant while she or her partner are participating in this study and for 3 months after study participation, the patient should inform the treating physician immediately
* Women of childbearing potential are required to have a negative serum pregnancy test (with a sensitivity of at least 25 mIU/mL) within 10-14 days and within 24 hours prior to the first dose of RO4929097 (serum or urine); a pregnancy test (serum) will be administered every 4 weeks if their menstrual cycles are regular or every 2 weeks if their cycles are irregular while on study; prior to dispensing RO4929097, the investigator must confirm and document the patient's use of two contraceptive methods, dates of negative pregnancy test, and confirm the patient's understanding of the potential of RO4929097 to cause serious or life-threatening birth defects; female patients of childbearing potential are defined as follows:

  * Patients with regular menses
  * Patients, after menarche with amenorrhea, irregular cycles, or using a contraceptive method that precludes withdrawal bleeding
  * Women who have had tubal ligation
* Female patients may be considered to NOT be of childbearing potential for the following reasons:

  * The patient has undergone total abdominal hysterectomy with bilateral salpingo-oophorectomy or bilateral oophorectomy
  * The patient is medically confirmed to be menopausal (no menstrual period) for 24 consecutive months
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients may not be receiving any other investigational agents
* Patients with known brain or leptomeningeal metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* Patients receiving any medications or substances that are inhibitors or inducers of CYP3A4 are ineligible
* Patients with malabsorption syndrome or other condition that would interfere with intestinal absorption; patients must be able to swallow tablets
* Known history of cirrhosis or clinically significant liver dysfunction
* Clinically significant hypocalcemia, hypomagnesemia or hypophosphatemia despite electrolyte supplementation
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia other than chronic, stable atrial fibrillation, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because RO4929097 is a Notch pathway inhibiting agent with the potential for serious or life-threatening birth defects or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with RO4929097, breastfeeding should be discontinued if the mother is treated with RO4929097; these potential risks may also apply to other agents used in this study
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with RO4929097; in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated
* Cardiovascular: baseline QTcF > 450 msec (male) or QTcF > 470 msec (female)
* Patients who have not recovered to < CTCAE grade 2 toxicities related to prior therapy are not eligible to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2010-05; Primary Completion 2011-05 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Strosberg, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with metastatic colorectal cancer who had received at least two prior lines of systemic chemotherapy were enrolled on the study.
Groups:
- Investigational Drug Therapy: RO4929097 20 mg by mouth 3 days on 4 days off continuously.
Period: Overall Study
Arm/Group | Investigational Drug Therapy
Started | 37
Completed | 33
Not Completed | 4
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Arm/Group | Investigational Drug Therapy
Number analyzed (Participants) | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 9
Age, Customized [Median (Full Range); unit: years] | 60 [42 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 22
Region of Enrollment [Number; unit: participants]
  United States | 37

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Objective Radiographic Response (ORR)
Description: To determine the objective radiographic response rate associated with RO4929097 in patients with metastatic colorectal cancer who have progressed following at least 2 prior treatments in the metastatic setting. Radiologic assessment of tumor burden (CT scans of the chest, abdomen and pelvis, or MRI of the abdomen and pelvis and CT of the chest) was scheduled every 8 weeks. Response Evaluation Criteria in Solid Tumors (RECIST version 1.1) were used for evaluation of the primary endpoint.
Time Frame: 2 months from enrollment for each participant
Population: All evaluable participants
Measure: Number; unit: participants
Arm/Group | Investigational Drug Therapy
Number analyzed (Participants) | 33
participants | 0

2. Secondary Outcome: Participant Overall Survival (OS) Rate
Description: Overall Survival defined as the time from start of treatment until death as a result of any cause, with patients censored at the date of last follow-up if still alive. The Kaplan-Meier method was used to estimate all time-to-event functions. Statistical analysis was performed using Stata SE 9.0 software and SAS 9.2 software.
Time Frame: Study duration of 12 months
Population: All evaluable participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Investigational Drug Therapy
Number analyzed (Participants) | 33
months | 6 [3.9 to 9.1]

3. Secondary Outcome: Participant Progression Free Survival (PFS) Rate
Description: Progression-Free Survival defined as the time from start of treatment until disease progression or death as a result of any cause. Patients were re-evaluated for response every 8 weeks. Response and progression were evaluated using the new international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1) [Eur J Ca 45:228-247, 2009]. Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes are used in the RECIST criteria.
Time Frame: Study duration of 12 months
Population: All evaluable participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Investigational Drug Therapy
Number analyzed (Participants) | 33
months | 1.8 [1.8 to 1.86]

4. Secondary Outcome: Number of Related Serious Adverse Events (SAEs)
Description: Study drug related grade 3-4 toxicities. To measure Adverse Events, investigators used the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Time Frame: Study duration of 12 months
Population: All evaluable participants
Measure: Number; unit: events
Arm/Group | Investigational Drug Therapy
Number analyzed (Participants) | 33
events | 0

ADVERSE EVENTS:
Time Frame: 12 months
Description: The toxicities considered possibly related to treatment are designated as such in the events listed below.
Arm/Group | Investigational Drug Therapy
Serious Adverse Events (participants affected / at risk) | 12/33
Other Adverse Events (participants affected / at risk) | 29/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational Drug Therapy (N=33)
Abdominal pain - unrelated (Gastrointestinal disorders) | 1 (1)
Anorexia - unrelated (Metabolism and nutrition disorders) | 1 (1)
Constipation - unrelated (Gastrointestinal disorders) | 1 (1)
Death - unrelated (General disorders) | 8 (8)
Dehydration - unrelated (Metabolism and nutrition disorders) | 1 (1)
Eye disorder - unrelated (Eye disorders) | 1 (1)
Headache - unrelated (Nervous system disorders) | 1 (1)
Hepatic failure - unrelated (Hepatobiliary disorders) | 1 (1)
Hepatic infection - unrelated (Infections and infestations) | 1 (1)
Ileus - unrelated (Gastrointestinal disorders) | 1 (1)
Leukocytosis - unrelated (Blood and lymphatic system disorders) | 1 (1)
Nausea - unrelated (Gastrointestinal disorders) | 4 (4)
Platelet count decreased - unrelated (Investigations) | 1 (1)
Pleural effusion - unrelated (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis - unrelated (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rectal pain - unrelated (Gastrointestinal disorders) | 1 (1)
Renal and urinary disorders - unrelated (Renal and urinary disorders) | 1 (1)
Small intestinal obstruction - unrelated (Gastrointestinal disorders) | 1 (1)
Vomiting - unrelated (Gastrointestinal disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational Drug Therapy (N=33)
Abdominal pain - unrelated (Gastrointestinal disorders) | 7 (8)
Alkaline phosphatase increased - unrelated (Investigations) | 1 (2)
Anorexia - unrelated (Metabolism and nutrition disorders) | 10 (10)
Back pain - unrelated (Musculoskeletal and connective tissue disorders) | 4 (4)
Blood bilirubin increased - unrelated (Investigations) | 1 (1)
Bronchopulmonary hemorrhage - unrelated (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chills - unrelated (General disorders) | 2 (3)
Constipation - unrelated (Gastrointestinal disorders) | 4 (4)
Cough - unrelated (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Diarrhea - unrelated (Gastrointestinal disorders) | 2 (2)
Dizziness - possibly related (Nervous system disorders) | 1 (1)
Dizziness - unrelated (Nervous system disorders) | 2 (2)
Dry eye - unrelated (Eye disorders) | 1 (1)
Dysgeusia - unrelated (Nervous system disorders) | 1 (1)
Dyspnea - unrelated (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Fatigue - possibly related (General disorders) | 1 (1)
Fatigue - unrelated (General disorders) | 3 (3)
Fever - unrelated (General disorders) | 4 (6)
Gastroesophageal reflux disease - unrelated (Gastrointestinal disorders) | 1 (1)
Gastrointestinal pain - unrelated (Gastrointestinal disorders) | 1 (2)
Headache - unrelated (Nervous system disorders) | 5 (5)
Hot flashes - unrelated (Vascular disorders) | 1 (1)
Hypertension - unrelated (Vascular disorders) | 2 (2)
Hypoglycemia - unrelated (Metabolism and nutrition disorders) | 1 (1)
Infections and infestations - unrelated (Infections and infestations) | 1 (1)
Insomnia - unrelated (Psychiatric disorders) | 2 (2)
Lethargy - unrelated (Nervous system disorders) | 1 (1)
Mucositis oral - possibly related (Gastrointestinal disorders) | 1 (1)
Nausea - possibly related (Gastrointestinal disorders) | 3 (3)
Nausea - unrelated (Gastrointestinal disorders) | 9 (9)
Neck pain - unrelated (Musculoskeletal and connective tissue disorders) | 1 (1)
Neutrophil count decreased - unrelated (Investigations) | 1 (1)
Non-cardiac chest pain - unrelated (General disorders) | 2 (2)
Oral pain - unrelated (Gastrointestinal disorders) | 1 (1)
Pain - unrelated (General disorders) | 1 (1)
Pain in extremity - unrelated (Musculoskeletal and connective tissue disorders) | 2 (2)
Pelvic pain - unrelated (Reproductive system and breast disorders) | 1 (1)
Productive cough - unrelated (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus - possibly related (Skin and subcutaneous tissue disorders) | 2 (2)
Pruritus - unrelated (Skin and subcutaneous tissue disorders) | 1 (1)
Rash acneiform - possibly related (Skin and subcutaneous tissue disorders) | 1 (1)
Rectal hemorrhage - unrelated (Gastrointestinal disorders) | 1 (1)
Skin hyperpigmentation - possibly related (Skin and subcutaneous tissue disorders) | 1 (1)
Urine discoloration - unrelated (Renal and urinary disorders) | 1 (1)
Urine output decreased - unrelated (Investigations) | 1 (1)
Vomiting - possibly related (Gastrointestinal disorders) | 2 (2)
Vomiting - unrelated (Gastrointestinal disorders) | 9 (9)
Weight loss - unrelated (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less